CLINICAL TRIAL: NCT00134394
Title: Double-Blind, Placebo-Controlled, Bilateral Comparison of Topical Tacrolimus 0.1% vs. Placebo Ointment as Adjunctive Therapy for Patients With Moderate to Severe Psoriasis Who Are Candidates for or Poor Responders to Etanercept Therapy
Brief Title: Etanercept With Tacrolimus for Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5085
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Psoriasis
Keywords: psoriasis; tacrolimus; etanercept
MeSH Terms: conditions — Psoriasis | interventions — Etanercept; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Etanercept plus tacrolimus

SUMMARY:
The study is designed to evaluate the efficacy of etanercept 50 mg subcutaneously (SQ) weekly plus tacrolimus 0.1% topical ointment twice daily compared to etanercept 50 mg SQ weekly plus placebo ointment twice daily.

DETAILED DESCRIPTION:
The study is designed to evaluate the efficacy of etanercept 50 mg SQ weekly plus tacrolimus 0.1% topical ointment twice daily compared to etanercept 50 mg SQ weekly plus placebo ointment twice daily. Subjects will be either beginning etanercept therapy or already using a stable dose of etanercept when they begin to apply tacrolimus to half of their body and placebo ointment to the other half. The study is double blinded. Total duration of the study is 12 weeks.

ELIGIBILITY:
Inclusion Criteria

* Adults 18 years or older with moderate to severe psoriasis, who are candidates for systemic or phototherapy, with a baseline score of 6 or higher on the target lesion score, and a baseline score of 3 or higher on the Physician's Global Assessment, on each side of the body
* Patients who are already on a stable dose of etanercept for at least 2 months and have the above criteria
* Subjects must have target lesions on each side of the body that are at least 1.5 cm in diameter and roughly symmetrical in appearance and location

Exclusion Criteria

* Inability to understand consent or comply with study requirements
* Pregnancy or unwillingness to use adequate birth control method
* Lactation
* Psoriasis plus ultraviolet A (PUVA) or systemic therapy within the past 4 weeks (other than a stable dose of Enbrel for at least 2 months)
* Ultraviolet B (UVB) or topical therapy (other than over-the-counter moisturizers) within the past 2 weeks
* Active tuberculosis or other opportunistic infection
* Demyelinating disease
* Uncontrolled congestive heart failure
* Known allergy to or any contraindications to using topical tacrolimus or etanercept
* Lack of insurance coverage or inability/refusal to pay out of pocket for etanercept and standard of care laboratory tests and PPD/CXR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-02; Study Completion 2007-12

PRIMARY OUTCOMES:
Target lesion scoring (on a scale of 0-12) at week 12
The percentage of lesions having scores of < 2 in the topical tacrolimus and vehicle-treated sites will be assessed.

SECONDARY OUTCOMES:
Photography of target lesions
Quarter-body photography
Static Physician's Global Assessment (PGA) on each side of each subject's body

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Magliocco, MD, Principal Investigator — UMDNJ - RWJMS
Locations (1):
- UMDNJ Psoriasis Center of Excellence, New Brunswick, New Jersey, United States